CLINICAL TRIAL: NCT07124104
Title: The Effect of Positive Psychotherapy-Based Self-Compassion Training on Internalized Stigma, Loneliness, and Empathy Levels of Parents of Children With Special Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, MÜJDE KERKEZ, Assist. Prof. Dr, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0000-0002-6968-9454
Record Dates: First submitted 2025-07-28; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Parental Stress; Internalized Stigma; Psychological Distress; Loneliness

STUDY DESIGN:
Intervention Model Description: RANDOMYZE CONTROL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Compassion Training Group (Experimental): Participants in this group will receive self-compassion training based on positive psychotherapy principles.
  Interventions: Behavioral: Positive Psychotherapy-Based Self-Compassion Training
- Control Group (No Intervention): Participants in this group will not receive any intervention.

INTERVENTIONS:
Behavioral: Positive Psychotherapy-Based Self-Compassion Training — Participants in the experimental group will receive Positive Psychotherapy-Based Self-Compassion Training, while participants in the control group will not receive any intervention.
  Arms: Self-Compassion Training Group

SUMMARY:
Parenting becomes more complex when it comes to raising children with special needs, introducing additional challenges. Unlike traditional parenting, raising a child with special needs requires adapting to constantly changing demands based on the child's individual needs. Furthermore, parents of children with special needs are at a higher risk of experiencing psychological distress compared to parents of typically developing children. High levels of internalizing and externalizing problems observed in children have been reported to cause high levels of stress in parents. Parents often experience complex emotions when they learn that their child has a disability. A child's disability can place a significant emotional and social burden on parents. As parents become more concerned about both their own future and that of their children, they may experience a variety of negative emotions such as stress, anxiety, and depression, which can negatively impact their health. Children with special needs often have developmental disorders such as autism, attention deficit hyperactivity disorder (ADHD), cerebral palsy, and physical disabilities, as well as visual, hearing, speech, behavioral, motor, and cognitive dysfunctions. Children with special needs are defined as individuals who require additional assistance and support from education, health, medical, and social-environmental services. Compared to raising typically developing children, being a parent of a child with special needs can lead to difficulties in family functioning, increased parenting stress, and inconsistent parenting styles. Therefore, examining the extent of psychological distress among parents of children with special needs is critical for developing solutions, interventions, and approaches to support parents. Self-compassion can be defined as developing a conscious awareness of the pain, distress, and negative emotions experienced by an individual, and adopting a kind, understanding, and supportive attitude toward oneself.This concept involves accepting one's shortcomings and failures as a natural part of being human, rather than harshly judging oneself, and being tolerant towards oneself in this process. Self-compassion is an internal attitude that enables an individual to accept negative experiences with balanced awareness and cope constructively, rather than denying or over-identifying with them. Self-compassion plays a crucial role in coping with emotional difficulties, particularly stress, anxiety, and depression. Individuals who cultivate self-compassion are able to learn from their mistakes and achieve a healthier emotional balance . Findings from self-compassion-based studies conducted with parents of children with disabilities suggest that increased levels of self-compassion are positively associated with various psychological and emotional well-being. A study conducted on parents of children with special needs found that as self-compassion increases, parents' optimism levels also increase. Similarly, Sumiati reported that self-compassion has a negative relationship with burnout and that individuals use more positive coping strategies as self-compassion increases. Stigmatization is the exposure of individuals to negative and exclusionary attitudes by others because they fall outside of the norms considered normal by society. This concept was first theorized by American sociologist Erving Goffman Stigma negatively impacts an individual's social status, leading to discrimination in social interactions. Internalized stigma, on the other hand, occurs when an individual internalizes the stigmatizing views held by society and develops negative perceptions of themselves. This can shape an individual's emotions, thoughts, beliefs, and fears, leading them to perceive themselves as dangerous, inadequate, or lacking in social adaptation. The effects of internalized stigma on an individual can have serious negative health consequences by exacerbating disease symptoms or prolonging the healing process. Individuals exposed to stigma feel shame because of their illness.they may develop attitudes such as feeling inadequate and avoiding social environments. This process can lead to a perception of worthlessness, fear of rejection, hopelessness and loss of self-confidence in individuals, which can negatively affect their psychological and social well-being. It has been found that parents of children with special needs are exposed to stigma. Loneliness is a complex and painful emotion that is difficult to define and understand, which individuals feel when they are distanced from their personal and social environments

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Able to read and understand Turkish
* Having a child with special needs (e.g., diagnosed developmental, behavioral, or psychiatric condition)
* Not having participated in any self-compassion or positive psychotherapy-based training in the past 6 months

Exclusion Criteria:

* Inability to read or understand Turkish
* Not having a child with special needs
* Having previously participated in any training programs for parents of children with special needs
* Not participating in the post-test
* Withdrawal from the study
* Receiving a psychiatric diagnosis according to DSM-5

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Change in Internalized Stigma Levels | Baseline and 5 weeks after the intervention
  Measured using the Parental Internalized Stigma Scale for Mental Illness (ERHİDÖ). This 29-item, self-report instrument assesses internalized stigma in parents of children diagnosed with a mental illness. It includes five subscales: alienation, stereotype endorsement, perceived discrimination, social withdrawal, and resistance to stigma. Items are rated on a 4-point Likert scale. Higher scores indicate higher levels of internalized stigma.
  [Cronbach's alpha = 0.87 for total scale; subscales range: 0.69-0.81]
Change in Self-Compassion Levels | Baseline and 5 weeks after the intervention
  Measured using the Self-Compassion Scale (SCS) developed by Neff (2003a) and adapted to Turkish by Akın et al. (2007). The scale consists of 26 items and six subscales: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Responses are given on a 5-point Likert scale (1 = "Almost Never" to 5 = "Almost Always"). Higher scores indicate greater self-compassion.
  [Cronbach's alpha for subscales ranges: 0.72-0.80]
Change in Empathy Levels | Baseline and 5 weeks after the intervention
  Measured using the Toronto Empathy Questionnaire (TEQ), developed by Spreng et al. (2009) and adapted into Turkish by Totan et al. (2012). The Turkish version contains 13 items with responses on a 5-point Likert scale. Items 1, 3, 5, 7, 8, 9, 11, and 12 are reverse-coded. Total scores range from 13 to 65, with higher scores indicating higher empathy.
  [Cronbach's alpha = 0.79]
Change in Loneliness Levels | Baseline and 5 weeks after intervention
  Measured using the UCLA Loneliness Scale - 8 item version (ULS-8), developed by Hays and DiMatteo (1987), and validated in Turkish by Doğan et al. (2011). The scale includes 8 items rated on a 4-point Likert scale (1 = "Never" to 4 = "Always"). Higher scores indicate greater loneliness.
  [Cronbach's alpha = 0.80]

CONTACTS AND LOCATIONS:
Locations (1):
- Batman University, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only aggregated results from statistical analyses will be reported or published. No identifiable or individual-level data will be made available.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT07124104/ICF_000.pdf